CLINICAL TRIAL: NCT05939765
Title: Pharmacologic Treatment in Legal Offenders With Schizophrenia, a Prospective Observational Mirror Image Study
Status: Withdrawn | Type: Observational
Why Stopped: After screening, not enough participants fulfilled the inclusion criteria.
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Stephan T. Egger, Principal Investigator, Psychiatric University Hospital, Zurich
Other Study IDs: AiW-TlG
Record Dates: First submitted 2023-06-25; First posted 2023-07-11 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Pharmacologic Treatment; Forensic Treatment; Antipsychotics; Violent Behavior
MeSH Terms: conditions — Schizophrenia | interventions — Antipsychotic Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antipsychotic — Participants will undergo a systematic neuropsychiatric assessement at regular intervals. Any change in medication, together with aggressive or dysfunctional behaviour will be continually recorded. The time period prior to the change in medication will be classified as control, the time after as case; therefore each patient becomes his own control.

SUMMARY:
Considering the vulnerability of patients with schizophrenia in forensic treatment, we have designed a prospective-observational trial. The purpose of our study, notably its focus on selecting the appropriate medication, developing clinical profiles, and determining the grounds of clinical judgment, is relevant for treating patients with schizophrenia.

DETAILED DESCRIPTION:
Patients with a schizophrenia spectrum disorder who commit violent crimes appear to have some distinguishing characteristics. The current view is that crime committed in the course of a psychiatric illness, particularly schizophrenia, is treatable and preventable. Nonetheless, treatment options for this patient group are sparse. The evidence regarding the efficacy and safety of such treatments is practically nonexistent. In practice therapeutic options are limited to medication and even here there is only one antipsychotic (clozapine) which has The current view is that crime committed during a psychiatric illness, particularly schizophrenia, is treatable and preventable. Nonetheless, treatment options for this patient group are sparse. The evidence regarding the efficacy and safety of such treatments is practically nonexistent. In practice, therapeutic options are limited to medication; even here, almost no controlled clinical trials are investigating this issue.

In clinical practice, selecting specific psychopharmacological treatments for patients with schizophrenia showing violent or aggressive behavior is particularly demanding. The lack of evidence regarding treatments for this particular group is partly attributable to their dual vulnerability and the consequent restrictions on clinical and experimental trials. Paradoxically, the efforts to ensure the safety and rights of these patients put them at a disadvantage, as they have no access to evidence-based treatment for their condition. Therefore, at best, they experience limited or slow improvement in their condition or, at worst, receive potentially ineffective or deleterious treatment.

To address the lack of evidence regarding the efficacy and safety of antipsychotic treatment options for this particular population, the investigators have designed a prospective observational study with evaluation in a mirror image design. This reduces confounders at the level of a randomized controlled trial, allowing for robust statistical analysis.

ELIGIBILITY:
Inclusion criteria

* Participants are competent to give informed consent.
* Participants are between 18 and 65 years of age.
* Diagnosis of schizophrenia DSM-5
* Violent crime in the course of a psychotic episode.
* German language proficiency

Exclusion criteria

* Low intelligence
* Current neurological disorder
* Substance induced psychotic disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Center for Inpatient Forensic Therapy (ZSFT: Zentrum für Stationäre ForensischeTherapie [German]), which is part of the Clinic for Forensic Psychiatry of the Psychiatric Hospital of the University of Zurich is Switzerland's largest forensic psychiatric clinic specializing in the treatment of imprisoned patients suffering from psychiatric disorders.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Psychopathology | 4 weeks
  The Positive and Negative Syndrome Scale (PANSS) is a semi-structured interview designed to meas-ure the severity of psychopathology in patients with a psychotic disorder. The scale ranges from 30 to 210; higher scores mean greater psychopathology. Change from baseline in psychopathology on the PANSS.

SECONDARY OUTCOMES:
Aggression | 12 Months
  The Modified Overt Aggression Scale (MOAS) is a four-part behavior rating scale used to evaluate and document the frequency and severity of aggressive episodes. It ranges 0 to 100: higher scores mean more severe aggression. Aggression and aggressive behavior as assessed by the MOAS.
Craving | 4 weeks
  The Yale Craving Scale (YCS) is a psychometric scale for assessing smoking and drinking urges. Total scores range from 0 to 40, with higher scores indicating greater dependence. Change from baseline in craving on the YCS.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan T. Egger, MD, PhD, Principal Investigator — University of Zurich
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jabat M, Redlich Bossy M, Bausch Becker N, Keppeler HC, Machetanz L, Kirchebner J, Vetter S, Seifritz E, Egger ST. Capacity to give informed consent in patients with severe mental disorder in different treatment settings. Front Psychiatry. 2026 Jan 2;16:1709553. doi: 10.3389/fpsyt.2025.1709553. eCollection 2025. PMID 41551193